CLINICAL TRIAL: NCT01815333
Title: Clinical and Technical Feasibility of a Ultrasuperparamagnetic Nanoparticle Iron Oxide (USPIO)-Enhanced Magnetic Resonance Lymph Node Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-0926; NCI-2014-02435 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cancer of Lymph Node
Keywords: Cancer of Lymph Node; Magnetic resonance imaging; MRI; Ultrasuperparamagnetic nanoparticle iron oxide; USPIO; Feraheme; Ferumoxytole
MeSH Terms: interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Feraheme (Experimental): Magnetic resonance imaging (MRI) acquired prior to the injection of Feraheme® and repeated at approximately 48 hours and 72 hours from the time of injection (scan time). The scan time will be adjusted, as needed. The MRI scan prior to the Feraheme injection is the routine scan. The scans at 48 and 72 hours are investigational.
  Interventions: Drug: Feraheme; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Feraheme — 6 mg of iron/kg (maximum 510 mg/dose) injected at a rate of 1 ml/sec (30 mg/sec) or slower after initial MRI.
  Other Names: Ferumoxytole
Procedure: Magnetic Resonance Imaging (MRI) — MRI scan performed before Feraheme injection. After Feraheme injection, MRI scan performed 2 days later, and then again the following day.

SUMMARY:
The goal of this clinical research study is to learn if the drug Feraheme ® (ferumoxytole) helps researchers most clearly to "see" cancerous lymph nodes on an MRI scan. Researchers also want to learn if ferumoxytole may be used in liver imaging.

Ferumoxytole is designed to deliver iron to treat iron-deficiency anemia (low red blood cell counts) in patients with chronic kidney disease. In this study, it will be used as an MRI contrast. Contrasts are used by doctors in order to see MRI images more clearly.

DETAILED DESCRIPTION:
Study Participation:

If you are found to be eligible, during the following MRI scans, you will pass into a long, narrow tube scanner, which is open at both ends. You will have a total of 3 MRI scans.

You will have an MRI scan before you receive ferumoxytole as needed. This is the standard-of-care MRI scan. You will then receive ferumoxytole by vein. If you are scheduled to have an MRI scan of your abdomen, or if you have visible lymph nodes in the abdomen, you will stay in the MRI scanner an extra 30 minutes for liver imaging right after you receive your dose of ferumoxytole. This is a part of an investigational scan (Visit 1--Day 1)

You will then return for an MRI scan 2 days later (Visit 2--Day 2) and then again the following day (Visit 3--Day 3) to scan your lymph nodes. These are the investigational scans. The timing of the second and third scans may be changed based on the study doctor's decision.

Length of Study:

Your participation on this study will be over after the third MRI scan.

Additional Information:

The images collected as part of this study will not be included as part of your medical record. If any of the images and/or information from this study are used for publication, all identifiable information will be removed. The data will be stored for 5 years after the study data has been published.

This is an investigational study. Ferumoxytole is FDA approved and commercially available for the treatment of iron-deficiency anemia in patients with chronic kidney disease. Its use to help researchers "see" cancerous lymph nodes from an MRI scan is considered investigational.

Up to 18 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled at MDACC, Written consent
2. Measurable nodes on the recent cross sectional imaging (CT, MRI. US) or suspicious lymph nodes for metastasis
3. Requiring tissue diagnosis (FNA, core biopsy, surgical biopsy, surgical resection), or clinical follow-ups for at least 6 months.
4. Any and all primary disease sites in the abdomen and pelvis will be allowed

Exclusion Criteria:

1. Primary or secondary iron overload
2. Lactation or pregnant - women of child bearing potential will be excluded
3. Contraindications for MRI
4. Contraindication or allergy to Feraheme® (based on insert)
5. Clinically documented or risk of primary or secondary iron overloading (e.g. History of thalassemia, sickle cell anemia, hereditary hemochromatosis, multiple transfusions with any reason), anemia not caused by iron deficiency
6. Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haesun Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2013 to July 2019. Recruitment took place at the University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Feraheme
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Feraheme
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Signal Intensity (SI) Change of a Lymph Node Between the Pre- and Post- Contrast of the Feraheme Enhanced Magnetic Resonance Imaging (MRI)
Description: Signal intensity (SI) change of a lymph node between the pre- and post- contrast images observed subjectively at each time point. The degree of SI change at each time point compared each other subjectively and a time point showing the nodes best (greatest signal loss relative to that on pre-contrast images) identified (optimum scan time).
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Feraheme
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: from injection, over the course of scanning, up to 3 days
Arm/Group | Feraheme
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT01815333/Prot_SAP_000.pdf